CLINICAL TRIAL: NCT06339840
Title: The Impact of Lifestyle Intervention on Weight and Fertility in Obese Males
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yichun Guan，PhD, Director, Reproductive Medicine Center,The Third Affiliated hospital of Zhengzhou University. Secretary-General, Asia Pacific Fertility Preservation Society, Third Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-036-01
Record Dates: First submitted 2024-03-14; First posted 2024-04-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Obesity; Weight Loss; Male Fertility; Artificial Insemination; IVF-ET
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Based on the design of this clinical trial, blinding is not implement ed for participants and care providers. Blinding is only applied to outcome assessors and investigators. Outcome assessors are clinical staff members who are unaware of the group assignments, and data is collected directly from the medical records system by EDC data entry personnel for management (double-checking). Data analysts will directly extract information and data from the EDC database for statistical analysis. Blinding will be revealed upon completion of result analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-carbohydrate diet group (Experimental): During the 12-week intervention, the first 8 weeks constitute the weight loss phase, where a low-carbohydrate diet, combined with meal replacement and daily dietary intake, is employed. Lifestyle guidance is provided on a one-to-one basis, accompanied by monitoring through a mobile platform. The subsequent 4 weeks involve the transition phase, during which personalized dietary and lifestyle adjustments are made
  Interventions: Dietary Supplement: Low-carbohydrate diet group
- Health Education Group (Other): 12 weeks of one-on-one health promotion and mobile platform monitoring
  Interventions: Behavioral: Health Education Group

INTERVENTIONS:
Dietary Supplement: Low-carbohydrate diet group — During the initial 8-week weight loss phase, participants will adopt a low-carbohydrate dietary pattern (with carbohydrate energy ratio of 20-30%, protein energy ratio of 30-40%, and fat energy ratio of 40-45%), with a caloric intake approximately 75% of their usual daily intake, but not less than 1200 kcal. Throughout the intervention period, participants will receive a daily nutritionally balanced meal replacement for 8 weeks to substitute for staple foods and control carbohydrate intake. Nutritionists will reinforce interventions by setting health goals, providing health education, implementing dietary and exercise interventions, and monitoring through a combined approach using a mobile platform. During the subsequent 4-week transition phase, participants' diets will gradually transition to a balanced dietary pattern (with carbohydrate energy ratio of 45-60%, protein energy ratio of 20-30%, and fat energy ratio of 20-25%) under the guidance of nutritionists.
  Other Names: Intensive Intervention Group
  Arms: Low-carbohydrate diet group
Behavioral: Health Education Group — Upon enrollment, nutritionists will provide lifestyle guidance to patients, including personalized adjustments such as limiting total energy intake to <1600 kcal/day, adjusting macronutrient distribution to 45-55% for carbohydrates, 20-30% for fats, and 20-30% for protein. Participants are advised to accumulate at least 150 minutes of moderate-intensity aerobic exercise per week (achieving 50%-70% of maximum heart rate). At enrollment, nutritionists will educate participants on healthy lifestyle principles, train them on nutritional intervention tools, and assist in food selection for weight management planning. Throughout the intervention, nutritionists will conduct follow-ups with patients via phone or mobile platforms to monitor weekly dietary and exercise habits, weight changes, and address any participant concerns promptly.
  Arms: Health Education Group

SUMMARY:
Obesity, defined by WHO standards as having a body mass index (BMI) equal to or greater than 30 kg/m², affects approximately 800 million people worldwide. It is evident that obesity has become a serious public health issue, resulting in significant health burdens.

Previous systematic reviews have indicated an association between obesity and male factor infertility. In populations undergoing assisted reproductive technology (ART), some studies have shown a correlation between increased male BMI and adverse ART outcomes. Furthermore, the negative effects of obesity may also be transmitted to offspring through genetic and epigenetic changes in reproductive cell DNA, increasing their risk of obesity, metabolic diseases, or other chronic conditions.

Currently, there is a lack of data on the impact of weight loss in obese men on fertility, and it is unclear which nutritional pattern in lifestyle interventions can more effectively control weight, improve semen quality, and address related endocrine issues in obese men, thereby improving reproductive treatment outcomes.

Based on previous literature, we hypothesize that lifestyle interventions, particularly strict low-carbohydrate diets combined with lifestyle guidance, may offer greater health benefits for obese men. These benefits include effective weight loss, improvement in semen parameters, reproductive metabolic health, quality of life related to reproductive health, and the impact on reproductive treatment outcomes. This provides a basis for non-pharmacological intervention strategies and methods for the health of obese men.

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged 22-40 years.
2. BMI≥30 kg/m² (defined as obesity according to WHO standards).
3. Patients who are willing and able to provide informed consent and follow all study procedures, including ongoing visits to the Reproductive Center of the Third Affiliated Hospital of Zhengzhou University and undergoing relevant tests
4. Spouse aged 20-40 years, with menstrual regularity (menstrual cycle length of 21-35days, duration of 2-7days), with a BMI of 18.5≤BMI < 25 kg/m², planning for AIH or IVF treatment at our center due to male factor infertility.
5. Not participating in any other research projects currently or in the preceding three months.
6. Willing to allow offspring conceived through the study to participate in follow-up research.

Exclusion Criteria:

1. Male reproductive urinary system abnormalities: active urinary reproductive system infections; hypogonadism; hyperprolactinemia; excessive estrogen; cryptorchidism, etc.;
2. Acute and chronic diseases that may affect fertility: chronic systemic diseases; history of systemic cytotoxic therapy or pelvic radiotherapy; other acute diseases that may affect study results;
3. Digestive system and metabolic abnormalities: acute and chronic digestive system diseases affecting digestive absorption function; history of or current eating disorders; allergies to ingredients in meal replacement products; gout, kidney stones, or gallstones; history of weight loss surgery;
4. Unhealthy lifestyle habits: meeting at least one of the following conditions: heavy alcohol consumption, daily smoking, history of drug abuse, history of substance abuse;
5. Personal factors affecting trial participation: impaired capacity to fully consent to participation in the study; major mental disorders; occupations requiring intense physical exercise; current diets that may interfere with the dietary plans of this study; exclusion of current or past use of hormones or anti-obesity drugs, or the use of other medications that affect hormone levels, carbohydrate metabolism, or appetite.

Ages: 22 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight | Regular data collection between baseline and 12 weeks of weight loss intervention
  kilogram (kg)

SECONDARY OUTCOMES:
Semen parameter- Sperm concentration | Collected at baseline and until 12 weeks after weight loss intervention
  Concentration (in million sperm cells/ml)
Semen parameter- Sperm motility | Collected at baseline and until 12 weeks after weight loss intervention
  Sperm motility (%)
Semen parameter- Sperm morphology | Collected at baseline and until 12 weeks after weight loss intervention
  Morphology (%)
Semen parameter- Sperm DNA fragmentation index (DFI) | Collected at baseline and until 12 weeks after weight loss intervention
  DFI (%)
Semen parameter- Sperm progressive motility (PR) | Collected at baseline and until 12 weeks after weight loss intervention
  PR(%)
Semen parameter- Non-progressive motility (NP) | Collected at baseline and until 12 weeks after weight loss intervention
  NP(%)
Semen parameter- Immotility (IM) | Collected at baseline and until 12 weeks after weight loss intervention
  IM(%)
body mass index (BMI) | Regular data collection between baseline and 12 weeks of weight loss intervention
  Calculated ad weight (kg)/height(m)^2
Waist circumference | Regular data collection between baseline and 12 weeks of weight loss intervention
  Centimetre(cm)
Hip circumference | Regular data collection between baseline and 12 weeks of weight loss intervention
  Centimetre(cm)
Lean mass | Collected at baseline and until 12 weeks after weight loss intervention
  (g), Assessed by an Anthropometric Analyzer
Fat mass | Collected at baseline and until 12 weeks after weight loss intervention
  (g), Assessed by an Anthropometric Analyzer
Abdominal fat | Collected at baseline and until 12 weeks after weight loss intervention
  (g), Assessed by an Anthropometric Analyzer
Visceral fat | Collected at baseline and until 12 weeks after weight loss intervention
  (g), Assessed by an Anthropometric Analyzer
Blood pressure | Regular data collection between baseline and 12 weeks of weight loss intervention
  mmHg
Heart rate | Regular data collection between baseline and 12 weeks of weight loss intervention
  beats per minute
Lipid profile-triglycerides | Collected at baseline and until 12 weeks after weight loss intervention
Lipid profile-LDL | Collected at baseline and until 12 weeks after weight loss intervention
  low-density lipoprotein
Lipid profile-HDL | Collected at baseline and until 12 weeks after weight loss intervention
  high-density lipoprotein
Lipid profile-VLDL | Collected at baseline and until 12 weeks after weight loss intervention
  very-low-density lipoprotein
Lipid profile-total cholesterol | Collected at baseline and until 12 weeks after weight loss intervention
Glucose metabolism-fasting glucose | Collected at baseline and until 12 weeks after weight loss intervention
Glucose metabolism-OGTT | Collected at baseline and until 12 weeks after weight loss intervention
  Oral Glucose Tolerance Test
Glucose metabolism-insulin | Collected at baseline and until 12 weeks after weight loss intervention
Glucose metabolism-C-peptide | Collected at baseline and until 12 weeks after weight loss intervention
Glucose metabolism-HbA1c | Collected at baseline and until 12 weeks after weight loss intervention
Sex hormones | Collected at baseline and until 12 weeks after weight loss intervention
  Samples will be analyzed for total testosterone, free testosterone, luteinizing hormone(LH), follicle-stimulating hormone(FSH), pituitary prolactin(PRL) and anti-müllerian hormone(AMH)

OTHER OUTCOMES:
Adult background | Collected prior baseline
  Demographic information and medical background
Questionnaire - Adult physical activity | Collected at baseline and until 12 weeks after weight loss intervention
  Physical activity will be assessed by the International Physical Activity Questionnaire (IPAQ)
Questionnaire - Quality of life | Collected at baseline and until 12 weeks after weight loss intervention
  Quality of life will be assessed by the validated tool, Short form-36 (SF-36).
Questionnaire - Psychological condition | Collected at baseline and until 12 weeks after weight loss intervention
  Psychological condition will be assessed by the validated tool, Depression-Anxiety-Stress Scale (DASS-21)
Questionnaire - Sleep | Collected at baseline and until 12 weeks after weight loss intervention
  Sleep will be assessed by the validated tool, Pittsburgh sleep quality index questionnaire (PSQI).
Spouse's reproductive outcome - Methods of Fertilization | through study completion, an average of 6 months
  The information will be collected through follow-up telephone calls or clinic registration. In the case of non-natural conception, specific assisted reproductive methods should be recorded in the registration
Spouse's reproductive outcome - Time to pregnancy | through study completion, an average of 6 months
  Duration of time to conception defined from time point allowed to conceive to registration of pregnancy.
Spouse's reproductive outcome - Length of gestational age | Assessed at birth of offspring
  gestational weeks
Spouse's reproductive outcome - Medication use | Collected from initiation of labor until completed birth of offspring
  Medication use during labor
Spouse's reproductive outcome - Delivery mode | Collected at birth of offspring
  Delivery mode (rupture of membranes or premature contractions, vaginal, cesarean section, instrumental delivery, miscarriage and stillbirth)
Spouse's reproductive outcome - Pregnancy complications | through study completion, an average of 18 months
  Pregnancy complications e.g. miscarriage, abortion (induced and indication for abortion), hydramnios, gestational hypertension, preeclampsia, need for maternal corticosteroid treatment for fetal lung maturation, urinary tract infection).
Spouse's reproductive outcome - Obstetrics complications | Collected at birth of offspring
  Obstetrics complications (e.g. preterm prelabour rupture of the membranes, shoulder dystocia, birth trauma (perinatal rupture), postpartum hemorrhage, maternal infections, maternal hospitalization)
Fetal and offspring - Apgar score | Collected at birth of offspring
  Apgar score (0-10). The higher the score, the better health condition of the offspring
Fetal and offspring - body weight | through study completion, an average of 18 months
  Fetal body weight will be measured with ultrasound during pregnancy and offspring body weight will be measured using an electronic scale.
Fetal and offspring - Neonatal fat mass | Assessed at birth (strived <24 hours, but allow <48 hours)
  Skinfold thickness measurement, millimeters (mm).
Fetal and offspring - Birth defects/abnormalities | Collected at birth of offspring
Fetal and offspring - length | through study completion, an average of 18 months
  Centimetre(cm)
Fetal and offspring - abdominal circumference | through study completion, an average of 18 months
  Centimetre(cm)
Fetal and offspring - crown circumference | through study completion, an average of 18 months
  Centimetre(cm)
Fetal and offspring - Glucose metabolism | Collected at 6, 12 and 18 months after birth
  Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for glucose, insulin, C-peptide and HbA1c
Fetal and offspring - Lipid profile | Collected at 6, 12 and 18 months after birth
  Parents will be instructed that the offspring should not have eaten two hours prior to the assessment.Samples will be analysed for triglycerides, LDL, HDL, VLDL and total cholesterol.
Fetal and offspring - Offspring growth factors and hormones | Collected at 6, 12 and 18 months after birth
  Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for Insulin-like Growth Factor 1 (IGF-1) and growth hormone (GH).
Fetal and offspring - Cognitive development of offspring | Collected at 6, 12 and 18 months after birth.
  Offspring cognitive development will be assessed by a Habituation and Free Play Test.
Labs - Semen epigenetics marks | Collected at baseline and until 12 weeks after weight loss intervention
  Epigenetic profile based on array-measurements. Analysed for methylation changes.
Labs - Adult Epigenetics | Collected at baseline and until 12 weeks after weight loss intervention
  Epigenetics analyses from whole blood. Will be analysed for methylation changes. The indicators for epigenetic testing include DNA methylation levels, histone modifications, non-coding RNA expression, etc.
Labs - Cord blood - epigenetics | Collected at birth
  Cord blood will be drawn immediately after birth and analysed for epigenetic profile.
Labs - Cord tissue | Collected at birth
  A sample of cord tissue will be collected immediately after birth and analysed for epigenetic profile.
Labs - Placenta | Collected at birth
  Placenta weight (gram).
Labs - Placenta - biopsies | Collected at birth
  Eight biopsies will be collected, four on the maternal site and four on the fetal side - one in each quadrant. The samples will be analyzed for protein expression patterns, placental markers, metabolomics, proteomics, markers of inflammation, immune markers and exosomes.
Labs - Offspring urine | Collected at birth and at 1, 3, 6, 12 and 18 months of age
  Parents will be instructed to collect offspring's urine samples. Offspring urine will be analyzed for metabolomics
Labs - Offspring feces | Collected at birth and at 1, 3, 6, 12 and 18 months of age
  Parents will be instructed to collect offspring's urine samples. Offspring urine will be analyzed for metabolomics

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China